CLINICAL TRIAL: NCT03470779
Title: A Randomized Controlled Wait-list Pilot Study Examining the Feasibility and Impact of a Combined Psychotherapy and Physiotherapy Group Treatment Program for Survivors of Torture Incarcerated in an Adult Prison in Kurdistan, Iraq
Brief Title: Impact of Combined Psychotherapy and Physiotherapy Group Treatment Program for Survivors of Torture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jeff Hartman, Assistant professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00206726
Record Dates: First submitted 2018-03-13; First posted 2018-03-20 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Pain Syndrome; Disability Physical
MeSH Terms: conditions — Somatoform Disorders | interventions — Physical Therapy Modalities; Psychotherapy

STUDY DESIGN:
Intervention Model Description: The study design is a randomized, wait-list controlled pilot study. A parallel group study design will be used to compare a treatment group and a wait-list control group. This study design will be effective for addressing the gap in literature by examining both the initial treatment estimates related to health and functioning and the feasibility of performing a similar study on a larger scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Participants randomly assigned to the treatment group will participate in an interdisciplinary treatment program in which local Kurdish psychotherapists and physiotherapists provide a 10-week intervention program. Treatment will consist of group physiotherapy and group psychotherapy
  Interventions: Other: Physiotherapy; Other: Psychotherapy
- Wait-list group (No Intervention): Participants randomly assigned to the wait-list group will not receive treatment but will participate in outcome data collection for comparison purposes.

INTERVENTIONS:
Other: Physiotherapy — Treatment group participants will participate in weekly group physiotherapy and psychotherapy sessions as part of the standard program procedure.
  Arms: Treatment group
Other: Psychotherapy — Treatment group participants will participate in weekly group physiotherapy and psychotherapy sessions as part of the standard program procedure.
  Arms: Treatment group

SUMMARY:
The aim of this study is to assess the impact and feasibility of an interdisciplinary group treatment approach, involving psychotherapy and physiotherapy, with survivors of torture that are incarcerated in a prison in Kurdistan, Iraq. The primary aim is to develop initial estimates of treatment effects on symptoms and poor functioning consistent with centralized pain and post-traumatic stress disorder, anxiety, and/or depression. The secondary aim is to assess the feasibility of studying this interdisciplinary treatment program in which local Kurdish psychotherapists and physiotherapists provide a 10-week intervention in a prison, in the Kurdish Sorani language, and to Kurdish participants that present with mental health symptoms, physical complaints, and poor functioning

DETAILED DESCRIPTION:
The aim of this randomized wait-list controlled pilot study is to assess the impact and feasibility of an interdisciplinary group treatment approach, involving psychotherapy and physiotherapy, with survivors of torture that are incarcerated in a prison in Kurdistan, Iraq. The primary aim is to develop initial estimates of treatment effects on symptoms and poor functioning consistent with centralized pain and post-traumatic stress disorder, anxiety, and/or depression. It is hypothesized that participants in the study will present with statistically significant improvements in some to all measures of symptoms and function. The secondary aim is to assess the feasibility of studying this interdisciplinary treatment program in which local Kurdish psychotherapists and physiotherapists provide a 10-week intervention in a prison, in the Kurdish Sorani language, and to Kurdish participants that present with mental health symptoms, physical complaints, and poor functioning

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* Incarcerated in the reformatory where research is conducted
* Native speaker of Sorani, a Kurdish language
* History of torture is reported and documented during the psychotherapy intake
* Presents with symptoms consistent with post-traumatic stress disorder, anxiety, and/or depression evident by a total score of greater than or equal to 1.75 on Hopkins Symptoms Checklist-25 and/or by a total score greater than or equal to 2.5 on the Harvard Trauma Questionnaire Part 4
* Presents with symptoms consistent with centralized pain evident by a score of greater than or equal to 40 on the Central Sensitization Inventory Part A.

Exclusion Criteria:

* Reports he will not remain in the current reformatory for at least 6 months from the onset of the study
* Is unable to make the time commitment required to participate
* Presents with symptoms consistent with a psychiatric condition which makes participation in the study unsafe for himself or others, based on the evaluation by the treating psychotherapist
* Presents with a high risk to self or others which makes participation in the study unsafe for himself or others, based on evaluation by the treating psychotherapist
* Participation is deemed unsafe due to a severe medical condition previously diagnosed by a medical doctor and/or signs/symptoms consistent with a possible medical condition based on the evaluation by the treating physiotherapist, 6.) reports previously receiving treatment by Wchan
* Current substance abuse reported by participant or identified by treating psychotherapist
* Currently receiving mental health services and/or physiotherapy services from other organization
* Reports unresolvable conflict with participant/s enrolled in the study.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This program and study are being administered in an all-male reformatory. Thus, only men are being studied.
Enrollment: 30 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist-25 | 10 weeks
  The HSCL-25 is a 25-question symptom inventory which measures symptoms of anxiety and depression.

SECONDARY OUTCOMES:
Patient Specific Functional Scale | 10-weeks
  This useful questionnaire can be used to quantify activity limitation and measure functional outcome for patients with any orthopaedic condition.
Pittsburgh Sleep Quality Index | 10-weeks
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults.
Patient's Global Impression of Change Scale | 10-weeks
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment
General Self Efficacy Scale | 10-weeks
  The General Self-Efficacy Scale is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life.
Central Sensitization Inventory | 10-weeks
  This tool was published with the purpose of providing a single self-report instrument that identified symptoms associated with central sensitization and the quantified the degree of those symptoms.
Harvard Trauma Questionnaire Part 4 | 10 weeks
  The Harvard Trauma Questionnaire (HTQ) is a checklist that inquires about a variety of trauma events, as well as the emotional symptoms considered to be uniquely associated with trauma.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff A Hartman, DPT, MPH, Principal Investigator — Northwestern University
Locations (1):
- Sulaymaniyah Adult Male Reformatory, Sulaymaniyah, Kurdistan, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
Still in deliberation